CLINICAL TRIAL: NCT01517568
Title: A Single-Centre, Open Label Trial Investigating the Metabolites in Plasma, Urine and Faeces After a Single Subcutaneous Dose of [3H]-Liraglutide to Healthy Subjects
Brief Title: Metabolism and Excretion of Liraglutide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1699; 2006-002293-22 (EudraCT Number)
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide [3H]

INTERVENTIONS:
Drug: liraglutide [3H] — A single dose of 0.75 mg will be given as a subcutaneous injection
  Other Names: [3H]-liraglutide

SUMMARY:
This trial is conducted in Europe. The aim of this trial is characterise the metabolic profile of liraglutide in plasma, urine, and faeces after a single injection of [3H]-liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the Investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs, and blood and urinary laboratory assessments
* BMI (Boday Mass Index) of 20.0-27.0 kg/m^2, both inclusive

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the Investigator
* Impaired renal function
* Active hepatitis B or active hepatitis C
* Positive human immunodeficiency virus (HIV) antibodies
* Any clinically significant abnormal ECG, as judged by the Investigator
* Any clinically significant abnormal laboratory test results, as judged by the Investigator
* Acute infection or inflammation or other illness that may influence the metabolism and excretion pattern of the trial product, as judged by the Investigator
* Known or suspected allergy to trial product(s) or related products
* History of alcoholism or drug abuse or positive results in alcohol and drug screens
* Smoking of more than 5 cigarettes per day
* Habitual excessive consumption of methylxanthine-containing (theophylline, caffeine or theobromine) beverages and foods (coffee, tea, soft drinks such as red bull, cola, chocolate) as judged by the Investigator
* Excessive consumption of a diet deviating from a normal diet, as judged by the Investigator

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Profile and identity of the major metabolites of tritium labelled liraglutide in plasma, urine, and faeces
Total recovery of tritium, [3H]-liraglutide and metabolites in urine and faeces

SECONDARY OUTCOMES:
Area under the curve
Cmax, maximum concentration
tmax, time to reach Cmax
t½, terminal half-life
The distribution of [3H]-liraglutide in whole blood versus plasma
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] Malm-Erjefalt M, Bjornsdottir I, Vanggaard J, Helleberg H, Larsen U, Oosterhuis B, van Lier JJ, Zdravkovic M, Olsen AK. Metabolism and excretion of the once-daily human glucagon-like peptide-1 analog liraglutide in healthy male subjects and its in vitro degradation by dipeptidyl peptidase IV and neutral endopeptidase. Drug Metab Dispos. 2010 Nov;38(11):1944-53. doi: 10.1124/dmd.110.034066. Epub 2010 Aug 13. PMID 20709939
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com